CLINICAL TRIAL: NCT06540690
Title: Comparison of Palatal Wound Healing in Diabetic and Non-diabetic Patients: Controlled Clinical Trial and in Vitro Study
Brief Title: Comparison of Palatal Wound Healing in Diabetic and Non-diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UEPJMF 14
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-01

CONDITIONS: Palate; Wound; Wound Heal; Diabetes
Keywords: Periodontology; Wound healing; Controlled Clinical Trial; Diabetes
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Controlled clinical study, non-randomized, prospective, blinded, with a three-month follow-up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic (D) (Active Comparator): Palatal wound healing in diabetic patients
  Interventions: Procedure: Palatal Wound
- Control Group (CG) (Active Comparator): Palatal wound healing in normoglycemic patients
  Interventions: Procedure: Palatal Wound

INTERVENTIONS:
Procedure: Palatal Wound — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive 4.0 silk sutures.

SUMMARY:
This study aims to characterize and compare the closure of open wounds in the palatal mucosa of diabetic and non-diabetic patients, evaluate clinical, patient-centered and immunological parameters as well as wound microbiome composition.

DETAILED DESCRIPTION:
The use of autogenous grafts from the palate for the reconstruction of gingival tissues is considered the gold standard for various periodontal and peri-implant reconstructions. Given the current aging of the population, it is essential to understand the cellular mechanisms responsible for the repair response in oral tissues and how they are affected by systemic diseases, such as diabetes mellitus (DM). The objectives of the present study, conducted through a controlled clinical trial, are to characterize and compare the closure of open wounds in the palatal mucosa of diabetic and non-diabetic patients. This will be achieved through clinical analyses, patient-centered parameters, inflammatory biomarkers, and wound microbiome composition. To accomplish this, 50 patients will be divided into two groups: the Diabetic Group (D; n = 25), where diabetic patients will undergo surgery for mucogingival defect correction with the addition of a free gingival graft, and the Control Group (GC; n = 25), where normoglycemic patients will undergo surgery for mucogingival defect correction with the addition of a free gingival graft. The groups will be compared regarding clinical parameters, patient-centered measures, including remaining wound area, epithelialization, tissue thickness, immature wound area, tissue edema, early wound healing index, postoperative discomfort, quality of life, number of analgesics, and sensitivity of the operated area over a 3-month period. Furthermore, the wound biofilm will be described through microbiome analysis, and tissue, saliva, and wound exudate biomarkers will be characterized. Descriptive statistics will be expressed as mean ± standard deviation, clinical evaluations will be performed using repeated measures ANOVA, and patient-centered parameters will be assessed using the T-test. Finally, multiple linear regression and correlation tests will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 18 years, systemically healthy, with good oral hygiene, assessed by plaque index and gingival index less than 25% (Ainamo, Bay, 1975);
* Patients with no morphological or pathological conditions on the palatine donor area;
* Patients who present indication for extraction and ridge preservation;
* The tooth included in the study, as well as, the adjacent teeth do not present loss of periodontal insertion;
* Patients who agreed to and sign the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 118 - May, 2012, and Ethics and Code of Professional Conduct in Dentistry - 118/12).
* Patients diagnosed with type 2 diabetes for more than 5 years who are using oral hypoglycemic agents or insulin supplementation, with HbA1c levels ranging from ≥ 6.1% to 8.5%.
* Non-diabetic patients with HbA1c levels below 6.1%.

Exclusion Criteria:

* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers patients;
* Pregnant or lactating patients;
* Patients who had had periodontal surgery on the study area;
* Patients who presents opportunistic oral lesions, mainly colonized the palate region;
* Use of dental prosthesis with palatal cover;
* Thin palatal mucosa (~2.0mm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Open Wound Area (OWA) | baseline, 7, 14, 21 days after surgery
  For this, standardized photographs will be taken. As a reference, a scale will be used to measure this area. These photographs will be exported to image software (Image J - National Institute of Health -NIH, Bethesda, USA), the area of the wound will be measured in square millimeters (Dias et al. 2015)

SECONDARY OUTCOMES:
Tissue Thickness (TT) | baseline, 90 days after surgery
  An endodontic spacer (Dentsply-Maillefer Instruments S.A. - Switzerland) with a rubber cursor will be placed in contact with the area until the palatal bone is reached, without pressing the tissue. The distance between the tip of the spacer and the cursor will be measured using a digital caliper (Dias et al., 2015).
Epithelialization (E) | baseline, 7, 14, 21, 30 e 90 days after surgery
  The wound will be colored with Shirley's solution and the epithelialized area will be quantified in the Image J. program. Then, with the total wound area, the % epithelialization will be calculated (Ozcelik et al., 2008).
Early wound healing index (EWHI) | 7 and 14 days after surgery
  According to Fickl et al. 2014 any modification in wound healing will be evaluated in five different degrees:
  Complete wound closure with an absence of fibrin on the palate; Complete wound closure with the presence of a fibrin line on palate; Complete wound closure with the presence of a clot with fibrin on palate Incomplete wound closure with partial tissue necrosis on palate; Incomplete wound closure with total tissue necrosis on palate
Tissue Edema (TE) | 7 days
  Tissue edema will be evaluated with the score: 1 = absent; 2 = slight; 3 = moderate; or 4 = severe (Sanz-Moliner et, 2013).
Oral Health Impact Profile (OHIP) | 14 days
  Will be evaluated from a questionnaire with 14 questions based on 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological deficiency and social deficiency. The patient should respond to the questions within 14 days after the surgical procedure, performing a postoperative diary. For each question an answer must be given, represented in numbers, being: 0- Never; 1- Almost never; 2-Occasionally; 3-Quite frequent; 4-Very common; 5-I do not know (Tonetti MS et al. 2017)
Number of analgesics | 14 days
  Number of analgesics used during 14 days after the procedure will be reported at the same postoperative diary (Tonetti et al. 2017).
Patient Discomfort | 14 days
  By a visual analogic scale (VAS) of 100 mm to assess discomfort, patients will report pain diary during the 14 days after surgery. Scale extremes will be "no pain" to "extreme." (Tonetti et al. 2017).
Qualitative somatosensory testing (QualST) | 7, 14 days
  This analysis will evaluate somatosensorial profiles and pain conditions. For this, different stimulus will be performed on the wound and the following tests will be applied: (1) Touch stimulus will be applied with a swab by a single application for 1-2 sec in the wound; (2) Cold stimulus will be applied by a stainless steel dental spatula (kept cool in ice water, approximately 0 °C) with wound direct contact during 1-2 sec; (3) The pinprick stimulus will be performed with a periodontal probe with moderate force on the wound area for 1-2 s (Baad-Hansen et al, 2013) Patient will report hypersensitivity, hyposensitivity, or normosensitivity to touch, cold and painful stimulus.
Immunologic Analysis | baseline, 3, 7 days
  With the goal to obtain baseline data for this parameter, crevicular gingival fluid from the gingival area next to the donor area will be collected previous surgery. An absorbent paper (PerioPaper, Oraflow, Plainview, NY, EUA) will be placed at wound edges without pressure during 40s. Collects with blood contamination will be discarded. Samples will be stored into a sterilized Eppendorf containing 100 μL Phosphate Buffer Saline 0.05% Tween 2 (PBS) at - 80 C. Growth factors (VEGF and EGF), chemokines (MIP-1α, MCP-1α), and cytokines (IL1β, IL6, IL10, TNFα) levels will be determinate by the multiplex assay. Moreover, MMP-2, MMP-9, TIMP-1, TIMP-2 will be measured by the same commercial human commercial kit.
Microbiome Analysis | baseline, 7, 14, 21, 30 e 90 days after surgery
  The biofilm from the palatal region will be collected, and the samples will be stored in sterilized Eppendorf tubes containing 100 μL of Phosphate Buffer Saline 0.05% Tween 20 (PBS) at -80°C. Three laboratory steps will be performed for the evaluation of the palatal region's microbiome, which are as follows: (1) Bacterial DNA extraction; (2) PCR amplification of the 16S rRNA region; (3) Library preparation for sequencing - PCR targeting the V3-V4 region. Bacterial DNA extraction will be conducted using a specific kit (MasterPure Complete DNA and RNA Purification Kit - Biosearch Technologies), following the steps of cell lysis and DNA purification.
Tissue Analysis | baseline
  To do so, the tissue sample collected during the surgical stage will be immediately immersed in 10% formaldehyde fixative for a period of 24 hours at room temperature. After the fixation period, the sample will be washed three times with a PBS solution at room temperature and then stored in 70% ethanol at 4°C. Using multiplexed immunofluorescence imaging technology (co-detection by indexing CODEX), a tissue atlas of the repair process will be generated for both healthy and diabetic patients. Biomarkers will be analyzed to determine the inflammatory profile, cell types, cell-cell contacts, and cellular neighborhoods, following the manufacturer's instructions (Black, 2021).
Saliva Analysis | baseline, 7 days
  After the collection of 5 ml of saliva, the sample will be centrifuged at 2800 g for 20 minutes at 4 ºC. The supernatant will be separated from the pellet, and to each 1 mL of saliva, 100 uL of a protease inhibitor solution (SIGMAFAST, Sigma, St. Louis, MO, USA) will be added. The following markers will be quantified through ELISA tests: (1) Histatin-1 (MBS2022124 H1, MyBioSource, San Diego, CA, USA), (2) Epidermal Growth Factor (EGF; KHG0061; Invitrogen, Waltham, MA, USA), and (3) Vascular Endothelial Growth Factor (VEGF-A; BMS277-2, Invitrogen, Waltham, MA, USA).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - College of Dentistry - São José dos Campos, Sao Paulo State University, São José dos Campos, São Paulo
  - Mauro Pedrine Santamaria and Ana Carolina Ferreira Bonafe, São José dos Campos, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the end of the study after a direct request
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688
- [Background] Kamalathevan P, Ooi PS, Loo YL. Silk-Based Biomaterials in Cutaneous Wound Healing: A Systematic Review. Adv Skin Wound Care. 2018 Dec;31(12):565-573. doi: 10.1097/01.ASW.0000546233.35130.a9. PMID 30475285
- [Background] Black S, Phillips D, Hickey JW, Kennedy-Darling J, Venkataraaman VG, Samusik N, Goltsev Y, Schurch CM, Nolan GP. CODEX multiplexed tissue imaging with DNA-conjugated antibodies. Nat Protoc. 2021 Aug;16(8):3802-3835. doi: 10.1038/s41596-021-00556-8. Epub 2021 Jul 2. PMID 34215862
- [Background] Fickl S, Fischer KR, Jockel-Schneider Y, Stappert CF, Schlagenhauf U, Kebschull M. Early wound healing and patient morbidity after single-incision vs. trap-door graft harvesting from the palate--a clinical study. Clin Oral Investig. 2014 Dec;18(9):2213-9. doi: 10.1007/s00784-014-1204-7. Epub 2014 Feb 23. PMID 24562700